CLINICAL TRIAL: NCT02969759
Title: Bioenergetics and Protein Metabolism in Sporadic Amyotrophic Lateral Sclerosis
Acronym: Fibro-ALS
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2016/36
Record Dates: First submitted 2016-11-04; First posted 2016-11-21 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Sporadic Amyotrophic Lateral Sclerosis
Keywords: Bioenergetics; Protein Metabolism; Sporadic Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic lateral sclerosis 1

ARMS (2):
- Patients (Other): ALS defined by El Escorial Criteria.
  Interventions: Other: Skin Biopsy
- Controls (Other): Asymptomatic subjects with normal examination.
  Interventions: Other: Skin Biopsy

INTERVENTIONS:
Other: Skin Biopsy

SUMMARY:
INTRODUCTION: Amyotrophic Lateral Sclerosis (ALS) is a degenerative disease of the motor neurones of the brain and the spinal cord. The pathophysiological mechanisms of the disease remain unknown. The average age of onset of ALS is about 60 years old, and the mean survival of patients is about 2 years. The disease is responsible for a progressive paralysis leading to death from respiratory failure. The only treatment available is the Riluzole, with a very modest efficiency on the progression of the disease. ALS is the third neurodegenerative disease, affecting 6000 persons in France, 150 000 in the world. Among the protagonists involved in the occurrence of the disease, mitochondrial perturbations and protein accumulations seem to be central elements.

OBJECTIVES: To precise the implication of energy and protein metabolism in the sporadic forms of ALS, to identify potential biomarkers of the disease and to test new therapies.

METHODS: The investigators will study cell growth, bioenergetics, mitochondrial dynamics, free-radicals production, presence of cytoplasmic inclusions, cytoskeleton structure and stress response in primary skin fibroblasts obtained from sporadic ALS patients. The study will be conducted over a period of three years in 3 centres specialized respectively in motor neuron diseases, mitochondrial metabolism and neuronal cytoskeleton.

PROSPECTS: If the investigators achieve to identify differences between ALS fibroblasts and controls, the results will be key elements to reinforce the hypothesis of a systemic disease with an important metabolic participation, to better define ALS pathophysiological mechanisms, to find potential biomarkers and to test new therapies.

DETAILED DESCRIPTION:
The investigators will study fibroblasts derived from sporadic ALS patients.

Clinical parameters will be collected such as sex, age, age of onset, clinical presentation, electrophysiological an respiratory parameters, treatments.

Patients and controls derived fibroblasts will be amplified and cultivated from skin biopsies.

Primary fibroblast cell cultures will be derived from skin biopsies obtained from control subjects and from the patients after obtaining written consent. Amplifications will be performed, from passage 1 to 6, allowing the time for cell cryopreservation of 10 samples per cell line. All experiments will be conducted on cells with similar passage numbers, ranging from 6 to 25, to avoid artefacts due to senescence.

Cell growth of each line will be monitored with the IncuCyte ZOOM® system (Essen Biosciences), a microscope gantry that resides in a cell incubator, and a networked external controller hard drive that gathers and processes image data. Cell growth will be automatically calculated at each time point using the relative cell density (ratio of the occupied area to the total area of the acquired regions).

The respiratory parameters of the fibroblasts will be monitored precisely with an high resolution oxygraph (OROBOROS). Enzymatic activity of each complex of the mitochondrial respiratory chain will be measured by spectrometry, and the mitochondrial membrane potential will be studied with fluorescence microscopy (TMRM probe). The investigators will also study mitochondrial dynamics and the architecture of mitochondrial network with fluorescence microscopy and super-resolution microscopy (SRM, Roper). The production of free radicals will be estimated with probes sensitive to oxidative stress. Finally, a metabolomic study (mass spectrometry QTRAP LC/MS/MS 5500 ABSciex) will be performed to characterise precisely the metabolites in the cells and to assess their metabolic profile.

The investigators will search for protein inclusions (intermediate filaments, TDP43, FUS, ubiquitin) with immuno-fluorescence technics. Western Blots will be performed to study the protein metabolism. The architecture of the cytoskeleton will be analysed in SRM and fluorescence microscopy, and the investigators will try to transfect fibroblasts in order to express Neurofilaments and study the consequences on the cytoskeleton and protein metabolism.

The investigators will study the response of the cells to the stress (hypoxia SCI-tive Dual, starvation), and to senescence (high passage numbers).

ELIGIBILITY:
Inclusion criteria :

* a free signed an written consent
* aged between 18 and 80 years old
* ALS defined by El Escorial Criteria
* normal neurological examination

Exclusion criteria:

* comorbidity or treatment susceptible to impact on metabolism
* differential diagnosis suspected, early and late forms (<6 month > 3 years)
* ALS not defined by El Escorial Criteria
* withdrawal of consent to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Kinetics of fibroblast growth | 24 hours
  The growth rates of the fibroblast lines

SECONDARY OUTCOMES:
Mitochondrial metabolism | 24 hours
  the breath parameters of fibroblast will be precisely studied by oxygraphy, a method consisting in measuring the oxygen consumption rates of fibroblasts in different metabolic phases
Protéic metabolism | 24 hours
  The presence of intracytoplasmic inclusion of target protein will be sought.
stress in senescence answer | 24 hours
  the answer due to the stress of cell lines in hypoxia and nutritionnal lack will be studied.